CLINICAL TRIAL: NCT05377957
Title: Prospective Registration Of Patient Data and Quality of Life in Eye Melanoma Patients
Acronym: PROQEM
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Nanda Horeweg, Senior researcher, department of radiation oncology, Leiden University Medical Center
Other Study IDs: PROQEM
Record Dates: First submitted 2022-04-19; First posted 2022-05-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma; Quality of Life; Shared decision-making; Patient preferences; Brachytherapy; Proton therapy; Enucleation
MeSH Terms: conditions — Uveal Melanoma; Patient Preference | interventions — Tape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Brachytherapy: Uveal melanoma patients treated with Ruthenium-106 plaque brachytherapy
  Interventions: Other: Quality of life questionnaires
- Proton therapy: Uveal melanoma patients treated with proton therapy
  Interventions: Other: Quality of life questionnaires; Other: Discrete choice experiment; Other: Shared decision-making analysis; Other: Impact of side-effects analysis
- Enucleation: Uveal melanoma patients treated with enucleation
  Interventions: Other: Quality of life questionnaires; Other: Discrete choice experiment; Other: Shared decision-making analysis; Other: Impact of side-effects analysis

INTERVENTIONS:
Other: Quality of life questionnaires — Collection of patient-reported outcomes concerning general and health-related quality of life and impact of uveal melanoma diagnosis
  Other Names: EORTC-QLQ-C30; EORTC-QLQ-OPT30; EQ-5D-5L; Impact of events scale
Other: Discrete choice experiment — Assessment of patient preferences for outcomes of proton therapy and enucleation
  Other Names: DCE
  Groups: Enucleation; Proton therapy
Other: Shared decision-making analysis — Assessment of shared decision-making from the perspective of the patient (by questionnaire), physician (by questionnaire) and a neutral observer (by audiotape), combined with patient-reported satisfaction and regret of the treatment decision (by questionnaire)
  Other Names: Audiotape; iSHARE; Satisfaction with decision scale; Decision regret scale
  Groups: Enucleation; Proton therapy
Other: Impact of side-effects analysis — Assessment of the impact of side-effects by questionnaire
  Groups: Enucleation; Proton therapy

SUMMARY:
PROQEM is a prospective cohort study among patients diagnosed with uveal melanoma to assess quality of life before and in the first five years after treatment.

DETAILED DESCRIPTION:
PROQEM is a prospective observational cohort study wherein patients with uveal melanoma are registered at diagnosis and are requested to fill in an array of questionaires before treatment and at 3, 6, 12, 24, 36 and 60 months after treatment. A comprehensive overview of the impact of their disease and treatment on quality of life is obtained by systematic assessment of the psychological impact of the initial diagnosis, eye symptoms, physical, emotional, social and role functioning.

In addition, the PROQEM has a substudy called the PROQEM-pco (Preferences, Choices and Outcomes) for the subgroup of patients who are eligible for both proton therapy and enucleation. They are invited to participate in research on patient preferences and shared decision-making. The consultations wherein the treatment decision is made are audiotaped and data on perceived shared decision-making, preferences, decision satisfaction and -regret are collected by questionaires at baseline and in the first 36 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical or pathological diagnosis of a melanoma of the choroid or ciliary body
* No signs of metastasis after staging procedures with at least an X-thorax, blood test and an ultrasound of the liver
* Treatment by brachytherapy, proton therapy or enucleation

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with uveal melanoma who will be treated with brachytherapy, proton therapy or enucleation with curative intent
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Uveal melanoma-related quality of life | 5 years
  EORTC QLQ-OPT30
Health-related quality of life | 5 years
  EORTC QLQ-C30
General quality of life | 5 years
  EQ-5D-5L
Impact of the diagnosis and treatment of uveal melanoma on mental health | 2 years
  Impact of events scale

SECONDARY OUTCOMES:
Patient preferences for outcomes of proton therapy and enucleation | Cross-sectional at baseline
  Discrete choice experiment
Shared decision-making | 1 year
  Audiotape, iSHARE, satisfaction with decision scale, decision regret scale
Impact of side-effects of treatment for uveal melanoma | 3 years
  Questionnaire specifically developed for uveal melanoma

CONTACTS AND LOCATIONS:
Overall Officials: Nanda Horeweg, Md PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The PROQEM study adheres to the FAIR principles of data stewardship. Due to privacy regulations the data of the PROQEM study will not be made publicly accessible, but can be made available upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After completion of the analysis and publication of the secondary endpoints by the PROQEM research group; until 15 years after the last publication.
Access Criteria: Data available upon reasonable request. A research proposal should be send to the chief investigator. Subject to ethical approval.